CLINICAL TRIAL: NCT03700762
Title: Application of Ultrasonic Gray-scale Ratio in Differentiating Benign From Malignant Thyroid Nodules.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-108-01
Record Dates: First submitted 2018-07-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Nodule; differential diagnosis
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — The patients will receive fine-needle aspiration of thyroid nodules after they have completed ultrasonic image tests. The cytological tests will be furtherly carried on in pathology department to confirm the histology of thyroid lesion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pathologically results: finally proved by pathologically results
- evaluate by ultrasound gray-scale ratio: the results confirmed by the cut-off value of ultrasound gray-scale ratio
  Interventions: Diagnostic Test: ultrasound gray-scale ratio

INTERVENTIONS:
Diagnostic Test: ultrasound gray-scale ratio — RADinfo radiograph reading system was used to measure the gray-scales of PTMC, NG, and thyroid tissues at the same gain level, the UGSR values of the PTMC, NG, and thyroid tissue were calculated.
  Groups: evaluate by ultrasound gray-scale ratio

SUMMARY:
According to the grades of echogenicity to evulated thyroid nodules is a subjective process and is thus influenced by the observer's judgement. The investigators first proposed the ultrasound gray-scale ratio (UGSR) to explore its efficacy for differentiating papillary thyroid microcarcinomas from small nodular goiters.

DETAILED DESCRIPTION:
Echogenicity is a common ultrasonic parameter to evaluate thyroid nodules. The echogenicity of the thyroid nodule was divided into 5 grades according to gray scale. Of the five categories, the diagnostic values of the hypoechoic and markedly hypoechoic categories have been widely accepted for thyroid malignant nodules. However, distinguishing between hypoechoic and markedly hypoechoic categories is a subjective process and is thus influenced by the observer's judgement. A more objective method should be proposed to differentiate papillary thyroid microcarcinoma(PTMC) from small nodular goiter(NG).

The investigators suspect the echo intensity of nodules could be reflected by values, as CT values reflecting the nodule density. The investigators first proposed the ultrasound gray-scale ratio (UGSR), namely, the ratio of lesion gray-scale value to surrounding normal thyroid tissue, and the previous study showed UGSR can better display the relationship of gray scale of PTMC or NG with surrounding normal thyroid tissue, and can make objective judgment of the nodules through quantitative results.

As the absolute ultrasound grayscale value is affected by the apparatus, scan gain, dynamic range, frequency, and operators. The investigators would collected different data acquired from different parameters to explore their potential relations.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as thyroid nodule.
* homo-echogenicity of normal thyroid tissue.
* able and willing to comply with all study requirements.

Exclusion Criteria:

* nodules are mainly cystic or calcified.
* pathology confirmed Hashimoto's thyroiditis.
* unable or unwilling to comply with all study requirements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with thyroid nodules by ultrasound or incidentally noted on other imaging tests.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic value of UGSR in differentiating benign from malignant thyroid nodules. | All the data will be uploaded in 1 year.
  The accuracy, sensitivity and specificity of UGSR in differentiating benign from malignant thyroid nodules.

SECONDARY OUTCOMES:
The best UGSR in differentiating benign from malignant thyroid nodules. | All the data will be uploaded in 1 year.
  The cut-off value of UGSR in differentiating benign from malignant thyroid nodules.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijiang Han, Doctor, Study Director — The Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine
Locations (1):
- The first people's hospital of Hangzhou, Hangzhou, Zhejiang, China